CLINICAL TRIAL: NCT04801953
Title: Intraoperative Application of Nimodipine to the Facial and Cochlear Nerves During Vestibular Schwannoma Resection to Avoid Spasm-related Postoperative Facial Paralysis and Deafness - a Prospective Randomized Pilot Study
Brief Title: Nimodipine in Vestibular Schwanommas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dorian Hirschmann, Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2263/2020
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nimodipine (Active Comparator): During surgery a nimodipine soaked gel foam pad is administered to the cranial nerves VII and VIII
  Interventions: Drug: NiMODipine Injectable Solution
- Placebo (Placebo Comparator): During surgery a sodium chloride soaked gel foam pad is administered to the cranial nerves VII and VIII
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NiMODipine Injectable Solution — nimodipine solution is applied to cranial nerves during resection of vestibular schwannoma
  Arms: Nimodipine
Other: Placebo — Sodium chloride solution is applied to cranial nerves during surgery
  Arms: Placebo

SUMMARY:
Title:

Intraoperative application of nimodipine to the facial and cochlear nerves during vestibular schwannoma resection to avoid spasm-related postoperative facial paralysis and deafness - a prospective randomized study

Background:

In patients undergoing microsurgical resection of a vestibular schwannoma, the facial and vestibulocochlear nerves are at risk. Prior studies suggested positive effects of nimodipine for preservation of the nerve function in these patients. A prospective, randomized, placebo controlled double-blinded study will be conducted to evaluate the neuro-protective effect of locally administered nimodipine during resection of vestibular schwannomas.

Investigational drug:

active group: "Nimotop® 10mg - Infusionsflasche" placebo: "Natrium chloratum physiologicum 0,9% - Medica Infusionslösung"

Rationale for the study: Nimodipine is supposed to counteract the vasoconstriction of cerebral arteries caused by microsurgical manipulation and might thereby preserve facial and cochlear nerve function

Aims of the study: Evaluation of the effect of intraoperative local administration of nimodipine on the postoperative function of the facial and vestibulocochlear nerves after microsurgical resection of vestibular schwannomas

Study design: prospective, double-blinded, single-center, randomized phase III trial

Study population: Patients undergoing microsurgical resection of a vestibularis schwannoma with a maximum diameter of 10-25mm on MRI at the Department of Neurosurgery, Medical university of Vienna.

Number of Patients: 30

Methods: In 15 patients, nimodipine will be administered locally to the facial and vestibulocochlear nerves during resection of a vestibular schwannoma (= treatment group). In another 15 patients, a placebo (sodium chloride solution) will be administered. In both cases, a soaked gel foam pad will be used. The operating team and the patient will both be blinded during the procedure. Facial nerve function and hearing will be assessed prior and three months after surgery.

Outcome variables: Serviceable or non-serviceable hearing according to Gardner-Robertson hearing scale and House-Brackmann score for the assessment of facial nerve function

Statistical analysis: For the evaluation of the postoperative function of the vestibulocochlear nerve, the number of patients with postoperative serviceable hearing (Gardner-Robertson I-II) and postoperative non-serviceable hearing (Gardner-Robertson III-V) will be compared between both groups. For the evaluation of the facial nerve function, the number of patients with favorable postoperative outcome (House-Brackmann I-III) and non-favorable postoperative outcome (House-Brackmann IV-VI) will be compared. In both cases, fisher's exact test will be used.

Expected risks/inconveniences: Administration of nimodipine is associated with the following adverse effects: thrombocytopenia, allergic reactions, headache, tachycardia, hypotension, nausea (occasionally) and bradycardia, ileus, reversibly elevated liver enzymes (seldom)

Risk/benefit assessment: Expected adverse effects of local nimodipine administration are manageable and patients may profit from the use of nimodipine. No severe adverse events are expected.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18a
* Vestibular schwannoma with maximum diameter of 10-25mm on MRI
* Pre-operative audiogram
* Informed consent

Exclusion Criteria:

* Contraindication for nimodipine application
* Vestibularis schwannoma diameter <10mm or >25mm on MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-04-09 (Estimated); Study Completion 2024-04-09 (Estimated)

PRIMARY OUTCOMES:
Facial nerve function | 90 days after surgery
  Function of the facial nerve according to House-Brackmann score. The House Brackmann score includes values from 1 to 6: 1 = normal function, 2 = minimal paresis, 3 = noticable paresis, 4 = severe paresis, 5 = minimum fuction, 6 = complete paralysis
Hearing | 90 days after surgery
  Serviceable or non-serviceable hearing according to Gardner-Robertson scale. The Gardner-Robertson scale indludes values from 1 to 5: 1 and 2 indicating serviceable hearing, 3-5 indicating non-serviceable hearing. The scores from 1 to 5 differ in values of pure tone audiometry and speech discrimination, 1 indicates best function and 5 worst function.

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Hirschmann, MD, Principal Investigator — University Clinic of Neurosurgery; Karl Roessler, MD, Principal Investigator — University Clinic of Neurosurgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No